CLINICAL TRIAL: NCT03344861
Title: A Multicenter, Prospective, Open-label, Non-randomized Single-arm Clinical Study of the Safety and Tissue Response to Photodynamic Therapy Using Porfimer Sodium for Injection as Treatment for Solid Lung Tumor Prior to Surgical Resection
Brief Title: Safety of PDT-Photofrin® Prior to Lung Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concordia Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI-PHO1701
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; Lung Cancer Metastatic
Keywords: lung cancer; lung carcinoma; lung metastases
MeSH Terms: conditions — Lung Neoplasms | interventions — Dihematoporphyrin Ether; Optical Fibers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Photodynamic therapy-Photofrin (Experimental): Photodynamic therapy (PDT) involves the i.v. injection of porfimer sodium (Photofrin®) followed by illumination of the tumor using a fiber optic device during navigational bronchoscopy. Two days after the injection, the laser light will be applied to the tumor.
  Interventions: Drug: Porfimer Sodium; Device: Fiber optic

INTERVENTIONS:
Drug: Porfimer Sodium — Porfimer sodium (Photofrin®) will be injected intravenously at a dose of 2 mg/kg.
  Other Names: Photofrin
Device: Fiber optic — After injection of porfimer sodium (Photofrin®), a flexible bronchoscopy with navigation guidance will be performed to confirm the location and the size of the lesion with the use of radial probe endobronchial ultrasonography (REBUS). An optical fiber diffuser length matching the tumor length will be placed in the lesion or adjacent to the lesion under fluoroscopy guidance. After the placement of the optical fiber, the laser light will be applied at a dose of 200 J/cm of diffuser length.

SUMMARY:
This research study is being conducted to assess the safety of PDT in subjects with peripherally located malignant tumors in lung parenchyma prior to surgical resection. It will involve up to 10 sites in USA. Participation will last 4 months.

DETAILED DESCRIPTION:
Lung cancer accounts for almost one-third of cancer deaths. Cancer screening strategies have the potential to achieve a 20% reduction in death rates. Newly developed bronchoscopic technologies (such as navigational bronchoscopy) have been shown to enable physicians to safely reach lesions in peripheral regions of the lung and obtain diagnosis. This new technology may now potentially offer bronchoscopic therapeutic interventions, such as photodynamic therapy, to tumors that were previously unreachable due to their peripheral anatomic location.

Photodynamic therapy (PDT) uses a combination of a photosensitizing drug (a drug that is activated by light), called porfimer sodium (Photofrin®), and a light from a laser that emits no heat. This technique works to allow the medical doctor to specifically target and destroy abnormal or cancer cells while limiting damage to surrounding healthy tissue. The activation of the drug is done by lightning the abnormal area using a fiber optic device (very fine fiber [like a fishing line] that permits light transmission) inserted into a flexible tube with a light, called bronchoscope for the lung. The light activates the porfimer sodium concentrated in the abnormal tissue, leading to its destruction.

The purpose of this study is to assess the safety of using photodynamic therapy prior to surgical resection of tumors located in the periphery of the lung.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-79
* Diagnosed with primary or metastatic tumor < 5 cm located in peripheral lung that can be completely resectable
* Candidate for surgical resection
* Candidate for bronchoscopy
* Tumor is accessible for unrestricted illumination of PDT
* Subject is deemed likely to survive for at least 3 months
* Non-menopausal/non-sterile female subject of childbearing potential has negative B-HCG (Human chorionic gonadotropin) at time of study entry
* Non-menopausal/non-sterile female subject of childbearing potential uses medically acceptable form of birth control
* Subject is able and willing to provide written informed consent to participate in the study, which must comply with ICH (International Council for Harmonisation) guidelines & local requirements

Exclusion Criteria:

* Diagnosis of small cell lung cancer or carcinoid tumors
* Primary or metastatic lung tumor located in central lung or near vertebral body
* Tumor invades a major blood vessel
* Presence of concurrent non-solid malignancy
* Tumor previously treated with radiation therapy
* Chemotherapy in the last four weeks
* Tumor treated with PDT within the last 3 months
* Abnormal blood results
* Subject with porphyria or hypersensitivity to Photofrin
* Coexisting ophthalmic disease likely to required slit-lamp exam within next 90 days
* Acute or chronic medical or psychological illness as judged clinical significant to PI to preclude bronchoscopy procedures
* female who is breast-feeding or intends to breast-feed during study
* subject who participated in another study within last 30 days or intends to participate in another study during this study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin O'Neil, Study Chair — Concordia Laboratories Inc.
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Cancer Treatment Centers of America/Southeastern, Atlanta, Georgia
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Dubois Medical Center, DuBois, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas
  - Providence Health & Services, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
This is a phase 2 study with only 10 subjects which is of minor use to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photodynamic Therapy-Photofrin
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Photofrin and Photodynamic Therapy: Open label study. All subjects had a 1-time administration of Photofrin and 1-time use of navigational bronchoscopy-PDT.
Arm/Group | Photofrin and Photodynamic Therapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Peripheral Lung Tumor [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With at Least One Adverse Event
Description: Safety evaluation will include incidence of all adverse events, including serious and non-serious. The count of how many subjects experienced at least one adverse event.
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 10
Statistical Analysis 1: Comparison: Photodynamic Therapy-Photofrin; Adverse events will be listed, coded by MedDRA, by system organ class and preferred term; Test type: Other — No comparator arm; p < 0.05, exact Clopper-Pearson binomial method; One-sided 95% upper confidence limit for the event percentage was calculated using exact (Clopper-Pearson) method for binomial proportion; Clopper-Pearson (binomial proportion) = .05 — One-sided 95% upper confidence limit for the event percentage was calculated using exact (Clopper-Pearson) method for binomial proportion

2. Secondary Outcome: Macroscopic Tissue Examination
Description: The mean measurement of tumor size after surgery. The largest diameter seen is measured.
Time Frame: Day 13 to 18
Population: Photodynamic therapy - Photofrin
Measure: Mean (Standard Deviation); unit: CM
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
CM | 2.177 (0.8003)

3. Secondary Outcome: Summary of Microscopic Tissue Examination: Percentage of Participants With Complete Response After Surgery
Description: The Percentage of Participants with Complete Response in Tumor area (no non-viable/necrotic tumor) after surgery
Time Frame: Day 13 to 18
Population: Look at complete response in the tumor area
Measure: Number; unit: percentage of participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
percentage of participants | 20

4. Secondary Outcome: Microscopic Tissue Examination: Percent Tumor Cell Necrosis in Tumor Area After Surgery
Description: The mean with standard deviation of the percent of tumor cell necrosis in the tumor area after surgery. The tumor itself was examined after it was removed to determine the percent of necrosis seen.
Time Frame: Day 13 to 18
Population: All subjects were examined for percent tumor cell necrosis in the tumor area
Measure: Mean (Standard Deviation); unit: Percent of tumor
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Percent of tumor | 22.0 (17.67)

5. Secondary Outcome: Microscopic Tissue Examination: Brisk Inflammatory Reaction After Surgery
Description: The number of participants showing a brisk inflammatory reaction in the tumor area after surgery. This is determined through a histological examination. Brisk Inflammatory Reaction is defined as lymphocytes that infiltrate diffusely the entire tumor and/or infiltrate across the entire base of the tumor.
Time Frame: Day 13 to 18
Population: The brisk inflammatory reaction percentage seen in the tumor area
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 9

6. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Cavitation in Normal Lung Area After Surgery
Description: The number of participants with cavitation seen in the normal lung area from the microscopic tissue examination after surgery
Time Frame: Day 13 to 18
Population: Number of participants with cavitation seen in normal lung area
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 1

7. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Hemorrhage Seen After Surgery
Description: The Number of Participants with hemorrhage seen during the microscopic tissue examination after surgery
Time Frame: Day 13 to 18
Population: Number of Participants with Hemorrhage seen in normal lung area after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 6

8. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Pneumonitis in the Normal Lung After Surgery
Description: The Number of Participants with pneumonitis seen in the normal lung area after surgery following the microscopic tissue examination
Time Frame: Day 13 to 18
Population: Microscopic Tissue Examination: Pneumonitis in the normal lung after surgery. Looked at Number of Participants with pneumonitis.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 2

9. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Increased Alveolar Macrophages in the Normal Lung After Surgery
Description: The number of participants with increased alveolar macrophages post surgery determined in the microscopic tissue examination.
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 10

10. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Atypical/Reactive Type 2 Pneumocytes in the Normal Lung After Surgery
Description: Number of Participants with Atypical/Reactive Type 2 pneumocytes seen in the normal lung after surgery during the Microscopic Tissue Examination:
Time Frame: Day 13 to 18
Population: Number of Participants with Atypical/Reactive Type 2 Pneumocytes in the normal lung after surgery determined during the Microscopic Tissue Examination.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 10

11. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Mucus Plugging/Mucositis in the Normal Lung After Surgery
Description: Number of Participants with Mucus Plugging/Mucositis seen in the normal lung after surgery during the Microscopic Tissue Examination.
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 0

12. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Interstitial Fibrosis in the Normal Lung After Surgery
Description: Number of participants with interstitial fibrosis in the normal lung after surgery seen during the Microscopic Tissue Examination
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  Mild | 0
  Moderate | 1
  Severe | 0
  None | 9

13. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Necrosis in the Normal Lung After Surgery
Description: Number of Participants with Necrosis seen in the normal lung after surgery during the Microscopic Tissue Examination
Time Frame: Day 13 to 18
Population: Number of Participants with Necrosis in the normal lung after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 3

14. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Large Vessel Damage Indicated by Fibrinoid Necrosis, Thrombus, Vasculitis in the Normal Lung After Surgery
Description: Number of Participants with Large Vessel Damage indicated by fibrinoid necrosis, thrombus, vasculitis in the normal lung after surgery seen during Microscopic Tissue Examination
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 1

15. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Acute Alveolar Damage in the Normal Lung After Surgery
Description: Number of Participants with Acute Alveolar damage in the normal lung after surgery seen during the Microscopic Tissue Examination
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 0

16. Secondary Outcome: Microscopic Tissue Examination: Number of Participants With Organizing Pneumonia Pattern in the Normal Lung After Surgery
Description: Number of Participants with Organizing pneumonia pattern in the normal lung after surgery seen during Microscopic Tissue Examination
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 7

17. Secondary Outcome: ECOG (Eastern Cooperative Oncology Group) Performance Status: Baseline
Description: Number of Participants with ECOG Performance at Baseline showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: Baseline (-30 to -1 Days)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 7
  ECOG 1 | 3

18. Secondary Outcome: ECOG Performance Status: Period 1 PDT Day 3
Description: Number of Participants with ECOG Performance Status at Period 1 PDT Day 3, showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 6
  ECOG 1 | 4

19. Secondary Outcome: ECOG Performance Status: Period II Surgery (Day 13-18)
Description: Number of Participants with ECOG Performance Status at Period II Surgery (Day 13-18) showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: Day 13 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 7
  ECOG 1 | 3

20. Secondary Outcome: ECOG Performance Status: Period III Follow-up (Day 20-25)
Description: Number of Participants with ECOG Performance Status at Period III Follow-up (Day 20-25) showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: Day 20 to 25
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 0
  ECOG 1 | 9
  ECOG 2 | 1

21. Secondary Outcome: ECOG Performance Status: Period III Follow-up (Day 43 -48)
Description: Number of Participants with ECOG Performance Status at Period III Follow-up (Day 43 -48) showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: Day 43 to 48
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 7
  ECOG 1 | 3

22. Secondary Outcome: ECOG Performance Status: Period III Follow-up (Day 103 - 108)
Description: Number of Participants with ECOG Performance Status at Period III Follow-up (Day 103 - 108) showing the number of participants at each ECOG level. ECOG is Eastern Cooperative Oncology Group. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  ECOG 0 | 9
  ECOG 1 | 1

23. Primary Outcome: Safety: Physical Examination Summaries of Non-normal Findings for Each Subject
Description: Safety evaluation will include the physical examinations summary of non-normal findings for each subject.
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  Respiratory abnormal at screening | 1
  Respiratory abnormal at Follow-up (Day 103-108) | 3
  Mouth abnormal at Follow-up (day 103-108) | 1

24. Primary Outcome: Safety: Vital Sign Summary of Abnormal Findings for Each Subject
Description: Safety evaluation will include vital sign summary for each subject. Only abnormal counts are included.
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 0

25. Primary Outcome: Safety: Laboratory Tests Summaries of Abnormal Findings for Each Subject
Description: Safety evaluation will include laboratory tests summarized for each subject with any abnormal lab results considered an AE (adverse event) to be listed.
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants
  Albumin (105-04) Period 1: 32 (drop of 10) | 1
  Lab values with no clinically significant change | 9

26. Primary Outcome: Safety: Skin Photosensitivity Events Summaries of Abnormal Findings for Each Subject
Description: Safety evaluation will include incidence of skin photosensitivity summarized for each subject.
Time Frame: 108 days (to 3 months post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 10
Participants | 4
Statistical Analysis 1: Comparison: Photodynamic Therapy-Photofrin; All adverse event terms are coded using MedDRA Dictionary version 21.1. NCS (Non-Clinical Significant) events were not included in the summary because their CTCAE grade and relationship were not collected. Subjects are counted once within each system organ class and each preferred term. An AE is defined as treatment related if its relationship to the study drug is recorded as "reasonable possibility" on the CRF (Case Report Form); Test type: Other; p < 0.05, exact Clopper-Pearson binomial method; One-sided 95% upper confidence limit for the event percentage, calculated using exact (Clopper-Pearson) method for binomial proportion

ADVERSE EVENTS:
Time Frame: Each subject was on study for 108 days. Study subjects were on study for 1 year 6 months in total (10Aug2017 to 7Feb2019).
Arm/Group | Photodynamic Therapy-Photofrin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy-Photofrin (N=10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) — On Study Day 4, subject received 2 doses of Toradol and on that same day complained of stomachache. On Study Days 4 & 5 subject had diarrhea. On Study Day 5 subject was diagnosed with moderate gastrointestinal bleed (CTCAE Grade 2).
Hemorrhagic Shock (Blood and lymphatic system disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced hemorrhagic shock (CTCAE Grade 4).
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced pleural effusion (recurrent right pleural effusion CTCAE Grade 2).
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced acute hypoxemic respiratory failure CTCAE Grade 4.
Anemia (Blood and lymphatic system disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced anemia CTCAE Grade 3.
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced iatrogenic right haemothorax CTCAE Grade 3 diagnosed from CT angiogram.
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced atrial fibrillation with rapid ventricular response CTCAE Grade 2 that converted to sinus.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject hospitalized for scheduled right colectomy for colon cancer and experienced dyspnoea CTCAE Grade 2.
Sepsis (Infections and infestations) | 1 (1) — Subject hospitalized with symptoms of cough, fever and chills resulting from sepsis CTCAE Grade 1.
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hospitalized with pneumonia aspiration CTCAE Grade 2 along with sepsis.
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — While hospitalized for sepsis and pneumonia aspiration, subject experience CTCAE Grade 2 SAE (Serious Adverse Event) of gastrooesophageal reflux disease
Deep Vein Thrombosis (DVT) Right (Blood and lymphatic system disorders) | 1 (1) — Hospitalized with CTCAE Grade 3 deep vein thrombosis right.
Deep Vein Thrombosis Left (Blood and lymphatic system disorders) | 1 (1) — While hospitalized with DVT Right, subject experienced a CTCAE Grade 2 SAE of deep vein thrombosis left.
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy-Photofrin (N=10)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) — Face swelling due to photosensitivity reaction.
Facial Blisters (Skin and subcutaneous tissue disorders) | 1 (1) — Blisters on face due to photosensitivity to drug.
Forearm Erythema (Skin and subcutaneous tissue disorders) | 2 (2) — Skin erythema on both forearms
Hand Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Mild hand erythema from photosensitivity to study drug.
Facial erythema (Skin and subcutaneous tissue disorders) | 2 (3) — Dermal erythema (sunburn) on face due to photosensitivity to study drug
Erythema on calves (Skin and subcutaneous tissue disorders) | 1 (1) — Dermal erythema (sunburn) on calves due to photosensitivity to study drug
Abdomen erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Abdomen redness due to photosensitivity to study drug.
Bradycardia (Cardiac disorders) | 2 (3)
Tachycardia (Cardiac disorders) | 1 (1)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (3)
Blood albumin decreased (Investigations) | 4 (4)
Blood alkaline phosphatase decreased (Investigations) | 1 (2)
Blood creatinine decreased (Investigations) | 2 (4)
Blood creatinine increased (Investigations) | 5 (7)
Blood glucose increased (Investigations) | 3 (6)
Blood pressure increased (Investigations) | 3 (8)
Blood pressure decreased (Investigations) | 1 (2)
Blood urea abnormal (Investigations) | 2 (3)
Blood urea increased (Investigations) | 1 (1)
Chest x-ray abnormal (Investigations) | 1 (2)
False negative investigation result (Investigations) | 3 (6)
Hematocrit decreased (Investigations) | 2 (2)
Hematocrit increased (Investigations) | 2 (2)
Hemoglobin decreased (Investigations) | 3 (4)
Hemoglobin increased (Investigations) | 2 (2)
Heart rate increased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
Prothrombin time abnormal (Investigations) | 2 (2)
Prothrombin time prolonged (Investigations) | 2 (2)
Red blood cell count decreased (Investigations) | 2 (2)
Red blood cell count increased (Investigations) | 1 (1)
Respiratory rate increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 2 (4)
x-ray abnormal (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2)
Protein deficiency (Metabolism and nutrition disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Respiratory abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Thoracic operation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 2 (6)
Hypotension (Vascular disorders) | 1 (2)
Blood Sodium increased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Prothrombin time shortened (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03344861/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03344861/SAP_001.pdf